CLINICAL TRIAL: NCT03622710
Title: Effects of Walking Training on Different Surfaces on Walking Ability, Balance Control, Lower Limb Muscle Strength, and Falls in Ambulatory Patients With Spinal Cord Injury
Brief Title: Effects of Walking Training on Different Surfaces on Walking Ability in Ambulatory Patients With Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Sugalya Amatachaya, School of Physical Therapy, Faculty of Associated Medical Sciences, Khon Kaen University, Khon Kaen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PHD57I0062
Record Dates: First submitted 2018-01-10; First posted 2018-08-09 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Spinal Cord Injuries; Rehabilitation
Keywords: Rehabilitation; Surfaces; Walking; Spinal cord injury
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Different surfaces (Experimental): Subjects are trained to walk over a walking track with different surfaces (WTDS) for 5 days over 4 weeks.
  Interventions: Other: Rehabilitation therapy
- overground (Active Comparator): Subjects are trained to walk overground for 5 days over 4 weeks.
  Interventions: Other: Rehabilitation therapy

INTERVENTIONS:
Other: Rehabilitation therapy — Subjects are trained to walk overground (control) or over WTDS (experimental) for 5 days/week over 4 week. Then they will be monthly follow-up for fall data.
  Other Names: Walking training

SUMMARY:
The study compares effects of 4-week walking training program on a walking track with difference surface [WTDS] and a firm ground on functional ability of ambulatory individuals with incomplete spinal cord injury [iSCI], using within- and between-group comparisons.

ELIGIBILITY:
Inclusion Criteria:

1. Age at least 18 years
2. Having an incomplete SCI (the American Spinal Cord Injury Association (ASIA) Impairment Scale or AIS C or D) (Kirshblum et al., 2011)
3. At a sub-acute or chronic stage of injury (post injury time: PIT > 3 months) (Wirth et al., 2008; Blackwell et al., 2001)
4. Able to walk with or without a walking device for at least 10m (Behrman et al., 2005; Lam et al., 2008; Jackson et al., 2008)
5. Having a body mass index (BMI) between 18.5-29.9 kg/m2 (Woo et al., 2007)

Exclusion Criteria:

1. Having an SCI from a progressive disease such as multiple sclerosis or malignancy
2. Having other medical conditions that might affect ambulatory ability, such as pain in the musculoskeletal system with an intensity of pain more than 5 out of 10 on a numeric rating pain scale (Dijkers, 2010), deformities of the spine and lower extremities (i.e. scoliosis, kyphosis, and equinovarus) and other neurological or other medical disorders (thromboembolism, autonomic dysreflexia).
3. Severe spasticity of the lower extremities (Modified Ashworth Scale (MAS) more than 2) (Bohannon & Smith, 1987; Scivoletto et al., 2008).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 72 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-07-15 (Actual); Study Completion 2019-01-16 (Actual)

PRIMARY OUTCOMES:
10-meter walk test (10MWT) | Change over 4 weeks
  Subjects walk at a comfortable pace along a 10m walkway. The test records the time use over the middle 4m of the walkway in order to minimize acceleration and deceleration effects. Then the average time over the 3 trials is converted to walking speed using the formula v=distance (m) /time (s)

SECONDARY OUTCOMES:
Timed up and go test (TUGT) | Change over 4 weeks
  Subjects stand up from a standard armchair, walk around a traffic cone that is located 3m away from the chair, and return to sit down on the chair at a maximum and safe speed. The test records the time taken from the command "Go" until the subject's back against the backrest of the chair. Then the average times finding over the 3 trials is used for data analysis.
Five times sit-to-stand test (FTSST) | Change over 4 weeks
  The time taken to complete 5 chair-rise cycles at a fastest and safe speed is measured for each subject. Then the average time over the 3 trials is used for data analysis.
6-minute walk test (6MWT) | Change over 4 weeks
  Subjects walk along a rectangular walkway as long as possible in 6 minutes. Every minute during the test, they are informed the time left and encouraged to continue in a good manner. Subjects are able to take a period of rest as needed and continued walking as soon as they can. The distance covered after 6 minutes are recorded
Incidence of fall | Six months after completing the training program.
  Then subject will be monthly monitored for the fall data during 6 months using a fall diary and telephone.

CONTACTS AND LOCATIONS:
Overall Officials: Sugalya Amatachaya, Principal Investigator — School of Physical Therapy, Faculty of Associated Medical Sciences, Khon Kaen University Affiliation: Khon Kaen University
Locations (1):
- Srinagarind hospital, Khon Kaen, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Amatachaya S, Promkeaw D, Arayawichanon P, Thaweewannakij T, Amatachaya P. Various Surfaces Benefited Functional Outcomes and Fall Incidence in Individuals With Spinal Cord Injury: A Randomized Controlled Trial With Prospective Data Follow-up. Arch Phys Med Rehabil. 2021 Jan;102(1):19-26. doi: 10.1016/j.apmr.2020.08.009. Epub 2020 Sep 11. PMID 32926851